CLINICAL TRIAL: NCT00741975
Title: Affect Management Intervention for Early Adolescents With Mental Health Problems
Brief Title: Affect Management Intervention for Early Adolescents Wtih Mental Health Problems
Acronym: Project TRAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH078750 (NIH); R34MH078750 (NIH)
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-02

CONDITIONS: HIV Infections
Keywords: HIV prevention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Affect Management
  Interventions: Behavioral: Affect Management
- 2 (Active Comparator): General Health Promotion
  Interventions: Behavioral: General Health Promotion

INTERVENTIONS:
Behavioral: Affect Management — 12-session group intervention including affect management training as well as sexual health skills training
  Arms: 1
Behavioral: General Health Promotion — 12-session group intervention including health information on a variety of developmentally relevant health topics
  Arms: 2

SUMMARY:
Adolescents are at risk for HIV because of sexual and drug use behavior initiated during early adolescence, and those with mental health problems appear to be particularly susceptible. Problems with managing emotions may make it difficult for early adolescents to make good decisions about sexual and substance use behaviors. This project will develop and evaluate interventions for early adolescents with mental health issues. An intervention focused on teaching affect management skills will be compared to an intervention addressing a variety of health topics to determine which intervention best reduces risk behavior among this at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Seventh graders identified by counselors at participating public school

Exclusion Criteria:

* Adolescent is HIV positive
* Adolescent is developmentally delayed
* Adolescent in pregnant
* Adolescent has a history of sexual crime

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2007-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Adolescent-reported sexual activity | 1 year

SECONDARY OUTCOMES:
Adolescent-reported condom use | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Houck, Phd, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States